CLINICAL TRIAL: NCT00527826
Title: A 12 Month Open-label Randomized Parallel Group Study to Investigate the Influence of Salmeterol Xinafoate/Fluticasone Propionate Either in Fixed Combination or Separately Via Diskus Inhalers on the Course of the Disease and Frequency of Exacerbations in Subjects With Severe and Very Severe COPD.
Brief Title: Influence Of Salmeterol Xinafoate/Fluticasone Propionate (50/500 µg BID) On The Course Of The Disease And Exacerbation Frequency In COPD Patients Gold Stage III And IV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCO107227
Record Dates: First submitted 2007-09-10; First posted 2007-09-11 (Estimated); Results first posted 2010-06-24 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Severe and very severe COPD (GOLD stage III / IV) exacerbations; health care utilisation; Chronic Obstructive Pulmonary Disease (COPD); quality of life; compliance; salmeterol/fluticasone combination
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Patient Compliance | interventions — Salmeterol Xinafoate; Fluticasone

ARMS (2):
- arm 1 (Active Comparator)
  Interventions: Drug: Salmeterol / Fluticasone (50/500 µg) BID fixed combination
- arm 2 (Active Comparator)
  Interventions: Drug: Salmeterol / Fluticasone (50/500 µg) BID separate Inhalers

INTERVENTIONS:
Drug: Salmeterol / Fluticasone (50/500 µg) BID fixed combination — comparator
  Arms: arm 1
Drug: Salmeterol / Fluticasone (50/500 µg) BID separate Inhalers — comparator
  Arms: arm 2

SUMMARY:
This is a 12 month randomized, open-label, parallel-group study to obtain data on the frequency and variability of exacerbations in severe and very severe Chronic Obstructive Pulmonary Disease (COPD) patients (Global Initiative for Chronic Obstructive Lung Disease (GOLD) Stage III and IV) receiving salmeterol xinafoate and fluticasone propionate either in fixed combination (SFC) or from separate inhalers (Sal/FP) with standard therapy. 200 subjects will be enrolled in approximately 30 study centres in Germany. Data on health care utilisation will be collected to compare direct costs associated with COPD in these two groups.

Baseline data will be collected for all subjects at Visit 1 and eligible subjects will be randomized to receive either SFC 50/500 µg bid (twice daily) as fixed combination or Sal 50 µg bid (twice daily) and FP 500 µg bid (twice daily) concurrently over 52 weeks. Subjects will return for study visits every two to three months until week 52. Additional telephone calls will be made between scheduled visits every 4 weeks. Assessments will include monitoring of frequency of exacerbations, health care utilisation (including emergency visits and hospitalizations) and rescue medication, lung function, drug compliance, health-related quality of life (SGRQ = St George's Respiratory Questionnaire) and safety.

DETAILED DESCRIPTION:
A 12 month open-label randomized parallel group study to investigate the influence of salmeterol xinafoate/fluticasone propionate either in fixed combination (SFC50/500 µg bid) or separately (SAL 50 µg and FP 500 µg bid) via Diskus inhalers on the course of the disease and frequency of exacerbations in subjects with severe and very severe COPD ( GOLD stage III+IV)

ELIGIBILITY:
Inclusion criteria:

* Subject must have a diagnosis of COPD based on the American Thoracic Society (ATS)/ European Respiratory Society (ERS) criteria.
* Male or female subjects, aged >=40 years. Females must be of Non Child Bearing Potential. The definition of Non Child Bearing Potential is as following: Females, regardless of their age, with functioning ovaries and who have a current documented tubal ligation or hysterectomy, or females who are post-menopausal.
* Have diagnosed COPD stage III or IV according to GOLD criteria: a baseline post-bronchodilator Forced Expiratory Volume, measured at 1 second (FEV1) <50% of predicted normal and a baseline post- bronchodilator FEV1/Inspiratory Vital Capacity (IVC) ratio <70%.
* Have experienced at least 2 moderate or severe COPD exacerbations leading to medical consultation (requiring oral corticosteroids or increasing dosage of oral corticosteroids and/or antibiotics or hospitalization) within the 12 months preceding Visit 1.
* Have stable COPD medication within 4 weeks prior to Visit 1 (no new medication added and no dosage changes in medication).
* Current or ex-smokers with a smoking history of at least 10 pack years (number of pack years = [number of cigarettes per day / 20] x number of years smoked, e.g., 20 cigarettes per day for 10 years, or 10 cigarettes per day for 20 years).
* Are currently managed at home (outpatients), are ambulatory and able to travel to the clinic. Subjects can be treated with all relevant COPD medication. This includes vaccines, inhaled short-acting beta-2-agonists as needed, short-acting or long-acting anticholinergics (tiotropium), systemic beta-2-agonists, theophylline, mucolytics, antioxidants, beta-1-agonists (for cardiovascular indication), non-invasive ventilation, long term oxygen therapy and can have Cor Pulmonale.
* A signed and dated written informed consent is obtained prior to participation.
* Able to comply with the requirements of the protocol and be available for study visits over 52 weeks.

Exclusion criteria:

* Known other respiratory disorders or signs for other respiratory disorders (e.g. asthma, lung cancer, sarcoidosis, tuberculosis, lung fibrosis, cystic fibrosis, bronchoectasis).
* Known history of significant inflammatory disease, other than COPD (e.g. rheumatoid arthritis and systemic lupus erythematosus).
* Known to be severely alpha-1-antitrypsin deficient (PI SZ or ZZ)
* Having undergone lung surgery (e.g. lung resection including lung volume reduction surgery, lung transplant) or subjects scheduled for surgery.
* Concurrent medication from Visit 1 and for the duration of the study with any of the prohibited medications: monoamine oxidase inhibitors and tricyclic antidepressants, and ritonavir (a highly potent cytochrome P450 3A4 inhibitor).
* Subjects receiving chronic or prophylactic antibiotic therapy.
* Serious, uncontrolled disease (including serious psychological disorders) likely to interfere with the study or impact on subject safety.
* Have, in the opinion of the investigator, evidence of alcohol, drug or solvent abuse.
* History of depression.
* History or presence of clinically significant drug sensitivity or clinically significant allergic reaction to corticosteroids or salmeterol.
* Moderate or severe COPD exacerbation (requiring corticosteroids or increased dosage of corticosteroids and/or antibiotics or hospitalization) within the 4 weeks prior to Visit 1
* Lower respiratory tract infection within the 4 weeks prior to Visit 1 .
* Pregnant or lactating female and female of childbearing potential.
* Subject is a participating investigator, sub-investigator, study coordinator, or other employee of a participating investigator, or is an immediate family member of the before mentioned. Subject is an employee of GlaxoSmithKline (GSK).
* Subject participated in an investigational drug study within 30 days prior to Visit 1

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2007-11; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (22):
- Germany (22):
  - GSK Investigational Site, Bruchsal, Baden-Wurttemberg
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Wiesloch, Baden-Wurttemberg
  - GSK Investigational Site, Cottbus, Brandenburg
  - GSK Investigational Site, Neuruppin, Brandenburg
  - GSK Investigational Site, Potsdam, Brandenburg
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Eschwege, Hesse
  - GSK Investigational Site, Gelnhausen, Hesse
  - GSK Investigational Site, Kassel, Hesse
  - GSK Investigational Site, Marburg, Hesse
  - GSK Investigational Site, Wiesbaden, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Gütersloh, North Rhine-Westphalia
  - GSK Investigational Site, Saarbrücken, Saarland
  - GSK Investigational Site, Annaberg, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Radebeul, Saxony
  - GSK Investigational Site, Berlin, State of Berlin
  - GSK Investigational Site, Schmölln, Thuringia

REFERENCES:
- [Derived] Hagedorn C, Kassner F, Banik N, Ntampakas P, Fielder K. Influence of salmeterol/fluticasone via single versus separate inhalers on exacerbations in severe/very severe COPD. Respir Med. 2013 Apr;107(4):542-9. doi: 10.1016/j.rmed.2012.12.020. Epub 2013 Jan 20. PMID 23337300

RESULTS

PARTICIPANT FLOW:
Groups:
- Salmeterol Xinafoate/FP in Fixed Combination (SFC) 50/500 µg: Salmeterol xinafoate/fluticasone propionate (FP) 50/500 µg twice a day (BID) (morning and evening) from the fixed combination inhaler (VIANI forte Diskus)
- Salmeterol Xinafoate/FP Separately (Sal/FP) 50/500 µg: Salmeterol xinafoate (Sal)/fluticasone propionate (FP) 50/500 µg BID (morning and evening) from two separate inhalers (SEREVENT Diskus and FLUTIDE forte Diskus)
Period: Overall Study
Arm/Group | Salmeterol Xinafoate/FP in Fixed Combination (SFC) 50/500 µg | Salmeterol Xinafoate/FP Separately (Sal/FP) 50/500 µg
Started | 108 (All Patients Population was used for Participant Flow section.) | 106
Completed | 87 | 80
Not Completed | 21 | 26
Not completed — Adverse Event | 10 | 10
Not completed — Lost to Follow-up | 3 | 2
Not completed — Withdrawal by Subject | 5 | 8
Not completed — Inclusion Criteria Not Met | 3 | 3
Not completed — Alpha-1 Antitrypsin Deficiency | 0 | 1
Not completed — Additional Intake of Viani forte | 0 | 1
Not completed — Participant moved away | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Salmeterol Xinafoate/FP in Fixed Combination (SFC) 50/500 µg | Salmeterol Xinafoate/FP Separately (Sal/FP) 50/500 µg | Total
Number analyzed (Participants) | 107 | 105 | 212
Age Continuous [Mean (Standard Deviation); unit: years] — Age at study start (years). The Intent-to-Treat (ITT) Population (all participants receiving at least one dose of study medication and suffering from COPD) was used for all baseline characteristics.
  years | 65.6 (8.3) | 64.2 (8.9) | 64.9 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants] — The ITT Population was used.
  Participants
    Female | 33 | 29 | 62
    Male | 74 | 76 | 150
Severity of Chronic Obstructive Lung Disease (COPD) [Number; unit: participants] — Severe COPD (stage III) is defined by the global initiative for chronic obstructive lung disease (GOLD) as baseline forced expiratory volume in one second (FEV1) >30% and <50% predicted and FEV1/inspiratory vital capacity (IVC) ratio <70%. Very severe COPD (stage IV) is defined as baseline FEV1 <30% predicted and FEV1/IVC <70%. ITT Population.
  participants
    Severe COPD | 77 | 79 | 156
    Very severe COPD | 30 | 26 | 56
Smoking History [Number; unit: participants] — The number of smokers/ex-smokers participating in the study was recorded. The ITT Population was used.
  participants
    Ex-smoker | 74 | 78 | 152
    Smoker | 33 | 27 | 60

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Exacerbations Per Year: Negative Binomial Model
Description: During regular visits, participants were asked whether they experienced any exacerbation since last contact. Between visits, COPD participants were contacted by phone by the staff and asked about exacerbation details. Exacerbations were defined according to Rodriguez-Roisin: moderate (grade II) exacerbations include a worsening of COPD symptoms that require both a change of respiratory medication (increased dose of prescribed or addition of new drugs) and medical assistance; severe (grade III) exacerbations include deterioration in COPD resulting in hospitalization or emergency room treatment.
Time Frame: Baseline through Week 52
Population: Intent-to-Treat (ITT) Population: all participants receiving at least one dose of study medication and suffering from COPD
Measure: Least Squares Mean (Standard Error); unit: Number of exacerbations per year
Arm/Group | Salmeterol Xinafoate/FP in Fixed Combination (SFC) 50/500 µg | Salmeterol Xinafoate/FP Separately (Sal/FP) 50/500 µg
Number analyzed (Participants) | 107 | 105
Number of exacerbations per year | 0.864 (0.134) | 0.862 (0.138)
Statistical Analysis 1: Comparison: Salmeterol Xinafoate/FP in Fixed Combination (SFC) 50/500 µg vs Salmeterol Xinafoate/FP Separately (Sal/FP) 50/500 µg; Test type: Non-Inferiority or Equivalence — Negative binomial model for the rate of exacerbations (per year) using the treatment duration as offset term and treatment, COPD severity (stratum) and interaction as fixed factors. This model took further into account a strata imbalance of 73% COPD III vs. 27% COPD IV according to the observed rates (SAS code: proc GENMOD); p = 0.73, Negative binomial model; Least square means adjusted for COPD severity (stratum), interaction of stratum with treatment, and strata imbalance of 73% COPD III vs. 27% COPD IV

2. Secondary Outcome: Compliance and Adherence to Study Medication
Description: Compliance is calculated as the ratio (in percent) between the number of actual doses taken during the total treatment period divided by the number of doses that should have been taken during the total treatment period.
Time Frame: Baseline through Week 52
Population: ITT Population
Measure: Mean (Standard Deviation); unit: percentage of doses
Groups:
- Sal 50 µg: Salmeterol xinafoate (Sal) 50 µg BID (morning and evening) from a separate inhaler (SEVERENT Diskus)
- FP 500 µg: Fluticasone propionate (FP) 500 µg BID (morning and evening) from a separate inhaler (FLUTIDE forte Diskus)
Arm/Group | Salmeterol Xinafoate/FP in Fixed Combination (SFC) 50/500 µg | Sal 50 µg | FP 500 µg
Number analyzed (Participants) | 107 | 105 | 105
percentage of doses | 97.08 (11.61) | 98.44 (19.62) | 98.33 (19.36)

3. Primary Outcome: Mean Number of Exacerbations Per Year: Poisson Model
Description: as for outcome 1
Time Frame: Baseline through Week 52
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Number of exacerbations per year
Arm/Group | Salmeterol Xinafoate/FP in Fixed Combination (SFC) 50/500 µg | Salmeterol Xinafoate/FP Separately (Sal/FP) 50/500 µg
Number analyzed (Participants) | 107 | 105
Number of exacerbations per year | 0.863 (0.136) | 0.830 (0.137)
Statistical Analysis 1: Comparison: Salmeterol Xinafoate/FP in Fixed Combination (SFC) 50/500 µg vs Salmeterol Xinafoate/FP Separately (Sal/FP) 50/500 µg; Test type: Non-Inferiority or Equivalence — Poisson model for the rate of exacerbations (per year) using the treatment duration as offset term and treatment, COPD severity (stratum) and interaction as fixed factors. This model took further into account a strata imbalance of 73% COPD III vs. 27% COPD IV according to the observed rates (SAS code: proc GENMOD); p = 0.66, Poisson model; [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: Mean Number of COPD-related Visits at/by Physician
Description: The total number of COPD-related visits, i.e., from baseline through week 52, the number of visits at physician's office, the number of home visits made by physician, the number of visits at an emergency outpatient clinic, as well as the number of home visits by an emergency physician were summed up.
Time Frame: Baseline through Week 52
Population: ITT Population with non-missing data (due to early withdrawal some data for this outcome measure are missing)
Measure: Mean (Standard Deviation); unit: number of visits
Groups:
- Total: Total number of participants randomized to the SFC and Sal/FP groups
Arm/Group | Salmeterol Xinafoate/FP in Fixed Combination (SFC) 50/500 µg | Salmeterol Xinafoate/FP Separately (Sal/FP) 50/500 µg | Total
Number analyzed (Participants) | 98 | 96 | 194
number of visits | 1.39 (2.33) | 1.06 (2.23) | 1.23 (2.28)

5. Secondary Outcome: Number of Participants With the Indicated Number of Days at the Intensive Care Unit (ICU)
Description: The number participants with the indicated number of days at the ICU was recorded.
Time Frame: Baseline through Week 52
Population: ITT Population of participants who were admitted to the ICU
Measure: Number; unit: participants
Arm/Group | Salmeterol Xinafoate/FP in Fixed Combination (SFC) 50/500 µg | Salmeterol Xinafoate/FP Separately (Sal/FP) 50/500 µg | Total
Number analyzed (Participants) | 25 | 16 | 41
participants
  0 days | 19 | 13 | 32
  1-5 days | 4 | 2 | 6
  6-10 days | 1 | 1 | 2
  11-30 days | 0 | 0 | 0
  >30 days | 1 | 0 | 1

6. Secondary Outcome: Number of Participants With the Indicated Number of Hospital Stays
Description: The number of participants with the indicated number of hospitalizations was recorded.
Time Frame: Baseline through Week 52
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Salmeterol Xinafoate/FP in Fixed Combination (SFC) 50/500 µg | Salmeterol Xinafoate/FP Separately (Sal/FP) 50/500 µg | Total
Number analyzed (Participants) | 107 | 105 | 212
participants
  0 hospital stays | 82 | 87 | 169
  1 hospital stay | 11 | 13 | 24
  2 hospital stays | 9 | 3 | 12
  3 hospital stays | 4 | 1 | 5
  4 hospital stays | 0 | 1 | 1
  5 or more hospital stays | 1 | 0 | 1

7. Secondary Outcome: Mean Number of Days Rescue Medication Was Used
Description: Participants were asked for the number of days they used rescue medication within the 7 days before Week 8 and Week 52.
Time Frame: The 7 days before baseline (=Visit 2 [Week 8]) and the last 7 days of study (=Visit 6 [Week 52])
Population: ITT Population with non-missing data (due to early withdrawal, some data for this outcome measure are missing).
Measure: Mean (Standard Deviation); unit: number of days
Arm/Group | Salmeterol Xinafoate/FP in Fixed Combination (SFC) 50/500 µg | Salmeterol Xinafoate/FP Separately (Sal/FP) 50/500 µg | Total
Number analyzed (Participants) | 101 | 98 | 199
number of days
  Visit 2 (Week 8) | 4.73 (2.37) | 4.11 (2.77) | 4.43 (2.58)
  Final visit (Week 52) | 5.03 (2.45) | 4.69 (2.67) | 4.86 (2.56)

8. Secondary Outcome: Mean Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) at Week 52
Description: Change from baseline was calculated as the FEV1 percent predicted value at Week 52 minus the percent predicted value at baseline. The post-bronchodilator lung function test was performed to measure FEV1 30 minutes after inhaling salbutamol. The most reliable result of three different consecutive measurements was documented.
Time Frame: Baseline and Week 52
Population: ITT Population
Measure: Mean (Standard Deviation); unit: percent of predicted value
Arm/Group | Salmeterol Xinafoate/FP in Fixed Combination (SFC) 50/500 µg | Salmeterol Xinafoate/FP Separately (Sal/FP) 50/500 µg | Total
Number analyzed (Participants) | 107 | 105 | 212
percent of predicted value
  Baseline | 36.82 (8.93) | 38.15 (9.26) | 37.47 (9.10)
  Week 52 | 38.98 (13.15) | 41.22 (15.26) | 40.09 (14.24)
  Mean change from baseline | 2.17 (10.42) | 3.08 (12.08) | 2.62 (11.26)

9. Secondary Outcome: Mean Change From Baseline in Inspiratory Vital Capacity (IVC) at Week 52
Description: Change from baseline was measured as the IVC value at Week 52 minus the value at baseline. The post-bronchodilator lung function test was performed to measure IVC 30 minutes after inhaling salbutamol. The most reliable result of three different, consecutive measurements was documented.
Time Frame: Baseline and Week 52
Population: ITT Population
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Salmeterol Xinafoate/FP in Fixed Combination (SFC) 50/500 µg | Salmeterol Xinafoate/FP Separately (Sal/FP) 50/500 µg | Total
Number analyzed (Participants) | 107 | 105 | 212
liters
  Baseline | 2.17 (0.74) | 2.29 (0.71) | 2.23 (0.72)
  Week 52 | 2.14 (0.72) | 2.27 (0.68) | 2.21 (0.70)
  Mean change from baseline | -0.02 (0.53) | -0.02 (0.50) | -0.02 (0.51)

10. Secondary Outcome: Mean Change From Baseline in the Tiffeaneau Index at Week 52
Description: The Tiffeneau index is defined as the FEV1 divided by the IVC (i.e., forced expiratory volume in one second relative to the inspiratory capacity) in percent. Change from baseline is calculated as the FEV1/IVC value at Week 52 minus the value at baseline.
Time Frame: Baseline and Week 52
Population: ITT Population
Measure: Mean (Standard Deviation); unit: percent of IVC
Arm/Group | Salmeterol Xinafoate/FP in Fixed Combination (SFC) 50/500 µg | Salmeterol Xinafoate/FP Separately (Sal/FP) 50/500 µg | Total
Number analyzed (Participants) | 107 | 105 | 212
percent of IVC
  Baseline | 48.90 (11.09) | 49.05 (10.76) | 48.98 (10.90)
  Week 52 | 50.82 (10.98) | 52.83 (16.39) | 51.81 (13.93)
  Mean change from baseline | 1.92 (8.76) | 3.78 (13.42) | 2.84 (11.32)

11. Secondary Outcome: Mean Change From Baseline in the Symptom Score of the St. George's Respiratory Questionnaire (SGRQ) at Week 52
Description: Change from baseline is calculated as the symptom score at Week 52 minus the symptom score at baseline. The SGRQ (a self-administered questionnaire) subscale symptom score ranges from 0 to 100% and measures the effect of respiratory symptoms, frequency, and severity on quality of life (summed weights of 8 questions). A score of 0 indicates the best possible status.
Time Frame: Baseline and Week 52
Population: ITT Population
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Salmeterol Xinafoate/FP in Fixed Combination (SFC) 50/500 µg | Salmeterol Xinafoate/FP Separately (Sal/FP) 50/500 µg | Total
Number analyzed (Participants) | 107 | 105 | 212
percent
  Baseline | 68.80 (19.65) | 68.95 (18.38) | 68.88 (18.99)
  Week 52 | 65.42 (19.76) | 63.77 (19.94) | 64.61 (19.82)
  Mean change from baseline | -3.38 (17.65) | -5.18 (17.27) | -4.27 (17.44)

12. Secondary Outcome: Mean Change From Baseline in the Activity Score of the St. George's Respiratory Questionnaire (SGRQ) at Week 52
Description: Change from baseline is calculated as the activity score at Week 52 minus the score at baseline. The SGRQ (a self-administered questionnaire) subscale activity score ranges from 0 to 100% and is concerned with activities that cause or are limited by breathlessness (summed weights of 2 questions). A score of 0 indicates the best possible status.
Time Frame: Baseline and Week 52
Population: ITT Population
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Salmeterol Xinafoate/FP in Fixed Combination (SFC) 50/500 µg | Salmeterol Xinafoate/FP Separately (Sal/FP) 50/500 µg | Total
Number analyzed (Participants) | 107 | 105 | 212
percent
  Baseline | 72.80 (17.78) | 70.64 (17.45) | 71.73 (17.61)
  Week 52 | 71.17 (20.29) | 68.53 (21.72) | 69.86 (21.01)
  Mean change from baseline | -1.63 (16.63) | -2.11 (16.53) | -1.87 (16.54)

13. Secondary Outcome: Mean Change From Baseline in the Impact Score of the St. George's Respiratory Questionnaire (SGRQ) at Week 52
Description: Change from baseline was calculated as the impact score at Week 52 minus the score at baseline. The SGRQ (a self-administered questionnaire) subscale impact score ranges from 0 to 100% and is concerned with social functioning and psychological disturbances (summed weights of 5 questions). A score of 0 indicates the best possible status.
Time Frame: Baseline and Week 52
Population: ITT Population
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Salmeterol Xinafoate/FP in Fixed Combination (SFC) 50/500 µg | Salmeterol Xinafoate/FP Separately (Sal/FP) 50/500 µg | Total
Number analyzed (Participants) | 107 | 105 | 112
percent
  Baseline | 46.03 (20.30) | 43.58 (17.37) | 44.82 (18.90)
  Week 52 | 44.66 (21.15) | 41.26 (19.53) | 42.98 (20.39)
  Mean change from baseline | -1.37 (17.52) | -2.32 (17.87) | -1.84 (17.66)

14. Secondary Outcome: Mean Change From Baseline in the Total Score of the St. George's Respiratory Questionnaire (SGRQ) at Week 52
Description: Change from baseline was calculated as the total score at Week 52 minus the score at baseline. The SGRQ (a self-administered questionnaire) total score ranges from 0 to 100% and summarizes the impact of COPD on overall health status (summed weights of 15 questions). A total score of 0 indicates the best possible status.
Time Frame: Baseline and Week 52
Population: ITT Population
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Salmeterol Xinafoate/FP in Fixed Combination (SFC) 50/500 µg | Salmeterol Xinafoate/FP Separately (Sal/FP) 50/500 µg | Total
Number analyzed (Participants) | 107 | 105 | 212
percent
  Baseline | 57.82 (17.07) | 55.89 (15.36) | 56.87 (16.24)
  Week 52 | 56.02 (18.22) | 53.25 (17.71) | 54.65 (17.98)
  Mean change from baseline | -1.80 (14.42) | -2.64 (14.73) | -2.22 (14.55)

15. Secondary Outcome: Mean Total Costs (Related to COPD) Per Participant
Description: Total costs include costs for hospitalization, medication, and visits to/by physician. Medications that were used "as required" were assumed to be used every second day.
Time Frame: Baseline through Week 52
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Euros per participant
Arm/Group | Salmeterol Xinafoate/FP in Fixed Combination (SFC) 50/500 µg | Salmeterol Xinafoate/FP Separately (Sal/FP) 50/500 µg | Total
Number analyzed (Participants) | 107 | 105 | 212
Euros per participant | 1453 (2427) | 1166 (1534) | 1311 (2034)

ADVERSE EVENTS:
Time Frame: Adverse events (AE) and serious adverse events (SAEs) were collected after the start of the study (visit 1, Week 0) until the last visit (visit 6, Week 52).
Description: The Safety Population (all participants who took at least one dose of study medication) was used for the analysis of SAEs/AEs. One participant in the Sal/FP group was excluded from the safety population because (s)he took no study medication (returned the study medication unused).
Arm/Group | Salmeterol Xinafoate/FP in Fixed Combination (SFC) 50/500 µg | Salmeterol Xinafoate/FP Separately (Sal/FP) 50/500 µg
Serious Adverse Events (participants affected / at risk) | 23/108 | 16/105
Other Adverse Events (participants affected / at risk) | 45/108 | 48/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Salmeterol Xinafoate/FP in Fixed Combination (SFC) 50/500 µg (N=108) | Salmeterol Xinafoate/FP Separately (Sal/FP) 50/500 µg (N=105)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 1
Cyanosis (Cardiac disorders) | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Duodenal stenosis (Gastrointestinal disorders) | 1 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 2 | 1
Pneumonia (Infections and infestations) | 3 | 4
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 12 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cardioplegia (Surgical and medical procedures) | 0 | 1
Arterial occlusive disease (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Salmeterol Xinafoate/FP in Fixed Combination (SFC) 50/500 µg (N=108) | Salmeterol Xinafoate/FP Separately (Sal/FP) 50/500 µg (N=105)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 33 | 33
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 12 | 16
Nasopharyngitis (Infections and infestations) | 3 | 8
Pneumonia (Infections and infestations) | 7 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.